CLINICAL TRIAL: NCT04324359
Title: A Multicenter, Randomized, Double-Masked Study To Compare The Ocular Safety, Tolerability, And Efficacy Of A Topical 0.2% Ophthalmic Corticosteroid Solution (SURF-201) To Vehicle In Cataract Surgery Subjects
Brief Title: Study to See How Well an Eye Drop, SURF-201, Works and What Side Effects There Are in Cataract Surgery Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Surface Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-201-001
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Post-surgical Ocular Inflammation; Post-surgical Ocular Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SURF-201 (Experimental): 0.2% topical preservative-free corticosteroid solution (0.2% betamethasone sodium phosphate)
  Interventions: Drug: SURF-201
- Vehicle (Placebo Comparator): Topical preservative-free vehicle (Placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SURF-201 — One drop twice daily (BID) in the study eye for 16 days.
  Other Names: 0.2% topical corticosteroid solution
  Arms: SURF-201
Drug: Placebo — One drop twice daily (BID) in the study eye for 16 days.
  Other Names: Vehicle
  Arms: Vehicle

SUMMARY:
SURF-201 is being studied for the treatment of eye inflammation and pain in people who are undergoing cataract surgery. SURF-201 is an investigational drug (which means the study drug is currently being tested) in the form of a sterile eye drop.

The purpose of this research study is to see how well SURF-201 works and what side effects there are, and to compare it with Vehicle (placebo). This study will involve about 80 study participants at several different research sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects age 18 years or older scheduled for uncomplicated unilateral cataract surgery with posterior chamber intraocular lens (IOL) implantation.
2. Subjects must be able to understand and sign the Informed Consent Form (ICF).
3. Female subjects of childbearing potential must agree to and submit a negative urine pregnancy test before any study-specific procedures are performed. The subjects must be using and continue to use a suitable method of contraception for the duration of the study: spermicide with barrier, oral contraceptive, transdermal contraceptive, injectable or implantable contraceptive, intrauterine device (IUD), abstinence or surgical sterilization of a partner. If a subject is not of childbearing potential (e.g., has been postmenopausal for at least 12 months or is premenarchal, or has undergone a hysterectomy, bilateral oophorectomy or a bilateral tubal ligation), a urine pregnancy test and use of a suitable method of contraception for the duration of the study will not be required.
4. Subjects must have a best-corrected visual acuity (BCVA) of at least +1.0 log of the minimum angle of resolution (logMAR) (Snellen equivalent of 20/200) in the non-study eye (fellow eye).
5. Subjects must have an intraocular pressure (IOP) of >8 mmHg and ≤22 mmHg in the study eye (surgery eye).
6. Subject must agree to maintain their current dosing regimen throughout the study period (from Screening through Day 32) if they are currently using topical cyclosporin-A or Xiidra (lifitegrast 5%).
7. Subjects must be willing and able to attend all study visits and follow all instructions.
8. Subjects must be able to self-instill the study drug (if unable, a caregiver must be available to instill all doses of the study drug).
9. Subjects must agree to avoid any medications which are disallowed (as defined by the protocol).

Exclusion Criteria:

1. Subject has any intraocular inflammation (cells and flare in the anterior chamber) or ocular pain (pain score of >0) in either eye prior to surgery.
2. Subject has any extraocular inflammation in the study eye prior to surgery (blepharitis is allowed if only scurf is present without any concurrent conjunctivitis or lid erythema/edema) or ongoing uveitis.
3. Subject has a history of diabetic retinopathy and/or previous vitrectomy in the study eye within the last 2 years prior to Screening which, in the investigator's opinion, is clinically significant and could impact the normal outcome of an uncomplicated cataract surgery.
4. Subject has a diagnosis of severe dry eye in the study eye.
5. Subject has any sign of iritis or scleritis in the study eye.
6. Subject has a history of glaucoma surgery in the study eye within the last 2 years prior to Screening.
7. Subject has a history of retinal surgery in the study eye within the last 2 years or plans to undergo retinal surgery in the study eye during the study period (from Screening through Day 32)
8. Subject has a history of Fuchs' dystrophy in the study eye.
9. Subject has guttata or chalazion in the study eye.
10. Subject has undergone radial keratotomy, photorefractive keratotomy, advanced surface ablation, corneal transplant, or LASIK in the study eye within the last 2 years prior to Screening.
11. Subject plans to undergo cataract surgery in the non-study (fellow) eye during the study period (from Screening through Day 32).
12. Subject plans to undergo additional ocular surgery (including femtosecond laser-assisted cataract surgery, minimally invasive glaucoma surgery, astigmatic keratotomy, limbal relaxing incision surgery, mechanical pupillary expanders, conjunctival incisions, and vitrectomy) in either eye during the study period (from Screening through Day 32).
13. Subject has a history of intraocular injections in the study eye within 6 months prior to Screening.
14. Subject has a history of herpes simplex infection in either eye.
15. Subject has active corneal, conjunctival or canalicular pathology (including ocular infection [bacterial, viral or fungal]) in the study eye. Specifically, active viral diseases of the cornea and conjunctiva including epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, and varicella, and also in mycobacterial infection of the eye and fungal diseases of the ocular structures (such as fungal keratitis).
16. Subject has thinning of the cornea or sclera.
17. Subject plans to undergo uncomplicated unilateral cataract surgery with the aid of anterior capsular staining products (e.g., Trypan blue) or with the aid of a femto (femtosecond) laser.
18. Subject has undergone anti-neoplastic therapy within the last 2 years prior to Screening or plans to undergo anti-neoplastic therapy during the study period.
19. Subject has a history of use of medications to treat benign prostatic hyperplasia that, in the opinion of the investigator, limits adequate dilation of the pupil to safely perform uncomplicated cataract removal and IOL implantation.
20. Subject has a history of liver disease within the last 5 years prior to Screening.
21. Subject has a history of previous ocular trauma in the study eye that places the study eye at risk of increased post-surgical complications or inflammation.
22. Subject has or had a known blood dyscrasia or bone marrow suppression.
23. Subject has an active or chronic/recurrent ocular or systemic disease that is not controlled and may have an impact on would healing (e.g., diabetes mellitus, systemic connective tissue disease, severe atopic disease).
24. Subject is suffering from alcohol and/or drug abuse.
25. Subject has a known hypersensitivity or poor tolerance to corticosteroids or any component of the study drug or any of the procedural medications such as anesthetic and/or fluorescein drops, dilating drops, etc.
26. Female subjects who are currently pregnant or nursing or are planning to become pregnant during the study or have a positive pregnancy test.
27. Subject has previously participated in this study protocol.
28. Subject used (within 30 days of initiation of study treatment) or is anticipating concurrent use of an investigational drug or device.
29. Subject has a condition or a situation which, in the investigator's opinion, might put the subject at increased risk, confound the study data or interfere significantly with the subject's study participation.
30. Subject would be wearing contact lens in either eye during the dosing period of Day -1 to Day 14.
31. Subject is taking a medication that the investigator feels might interfere with the study parameters.
32. Subject tests positive for the Coronavirus Disease 2019 (COVID-19) virus prior to Visit 1 (Day -14 to Day -2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Hosseini, MD, PhD, Study Chair — Surface Ophthalmics, Inc.
Locations (10):
- United States (10):
  - Inland Eye Specialists, Hemet, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Hernando Eye Institute, Brooksville, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Alterman, Modi & Wolter, Poughkeepsie, New York
  - Eye Care Specialists, Kingston, Pennsylvania
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Texan Eye Care, PA - Keystone Research, Ltd., Austin, Texas
  - R and R Eye Research, LLC, San Antonio, Texas

REFERENCES:
- [Background] Hosseini K, Gollamudi S, Reiser H, Walters T, Lindstrom RL. 0.2% Betamethasone Sodium Phosphate: A Multicenter, Randomized, Double-Masked Study to Compare Its Ocular Safety, Tolerability, and Efficacy to Vehicle in Cataract Surgery Subjects. Clin Ophthalmol. 2023 Aug 5;17:2219-2230. doi: 10.2147/OPTH.S419857. eCollection 2023. PMID 37564159
- See also: 0.2% Betamethasone Sodium Phosphate: A Multicenter, Randomized, Double-Masked Study to Compare Its Ocular Safety, Tolerability, and Efficacy to Vehicle in Cataract Surgery Subjects. — https://doi.org/10.2147/OPTH.S419857

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SURF-201 | Vehicle
Started | 40 | 43
Completed | 39 | 41
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Randomized participants who underwent routine uncomplicated cataract surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | SURF-201 | Vehicle | Total
Number analyzed (Participants) | 39 | 43 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (6.82) | 68.4 (9.90) | 68.4 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 12 | 18 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 36 | 38 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 31 | 33 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Anterior Chamber Cell (ACC) Grade at Baseline [Count of Participants; unit: Participants] — Number of participants with a baseline ACC Grade of 0 (i.e., no ACCs seen)
  Participants | 39 | 43 | 82
Ocular Pain Score at Baseline [Count of Participants; unit: Participants] — Number of participants with a baseline Ocular Pain Score of 0 (no pain)
  Participants | 39 | 43 | 82

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Cell (ACC) Grade: Number of Participants Achieving an ACC Grade of 0
Description: The Investigator used a slit lamp biomicroscope to assess ACCs in the study (surgery) eye. ACC counts were graded as follows:
  ACC Grade 0 = 0 cells were seen ACC Grade higher than 0 = 1 or more cells were seen
Time Frame: Day 15
Population: Randomized participants who had uncomplicated cataract surgery. Missing values were imputed using last observation carried forward (LOCF).
  LOCF is a common statistical approach to the analysis of longitudinal repeated measures where some follow-up (FU) observations may be missing. In a LOCF analysis, a missing FU value is replaced by (imputed as) that participant's previously observed value. The combination of the observed and imputed data is then analyzed as if there were no missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | SURF-201 | Vehicle
Number analyzed (Participants) | 39 | 43
Participants | 22 | 9
Statistical Analysis 1: Comparison: SURF-201 vs Vehicle; Test type: Superiority; p < 0.001, z-test for proportions; Other: z-test for proportions, 2-sided test at alpha = 5% level. P-value: based on the normal approximation test for differences between proportions

2. Secondary Outcome: Post-surgical Ocular Pain Score: Number of Participants Achieving an Ocular Pain Score of 0
Description: Ocular pain was assessed and graded by the participants using the Visual Analog Scale (VAS). The VAS was scored from 0 to 100 using a mark on the 100 mm line (0=absent [no pain], 100=maximum [severe pain]).
Time Frame: Day 1
Population: Randomized participants who underwent routine uncomplicated cataract surgery and had no missing assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | SURF-201 | Vehicle
Number analyzed (Participants) | 39 | 43
Participants | 27 | 21
Statistical Analysis 1: Comparison: SURF-201 vs Vehicle; Test type: Superiority; p = 0.066, Other: z-test for proportions; Other: z-test for proportions, 2-sided test at alpha = 5% level. P-value: based on Barnard's exact test for differences between proportions

3. Secondary Outcome: Post-surgical Ocular Pain Score: Number of Participants Achieving an Ocular Pain Score of 0
Description: as for outcome 2
Time Frame: Day 8
Population: Randomized participants who underwent routine uncomplicated cataract surgery and had no missing assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | SURF-201 | Vehicle
Number analyzed (Participants) | 39 | 41
Participants | 32 | 32
Statistical Analysis 1: Comparison: SURF-201 vs Vehicle; Test type: Superiority; p = 0.716, z-test for proportions; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Post-surgical Ocular Pain Score: Number of Participants Achieving an Ocular Pain Score of 0
Description: as for outcome 2
Time Frame: Day 15
Population: Randomized participants who underwent routine uncomplicated cataract surgery and had no missing assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | SURF-201 | Vehicle
Number analyzed (Participants) | 39 | 40
Participants | 35 | 33
Statistical Analysis 1: Comparison: SURF-201 vs Vehicle; Test type: Superiority; p = 0.528, z-test for proportions; Other: z-test for proportions, 2-sided test at alpha = 5% level P-value: based on Barnard's exact test for differences between proportions

5. Secondary Outcome: Post-surgical Ocular Pain Score: Number of Participants Achieving an Ocular Pain Score of 0
Description: as for outcome 2
Time Frame: Day 22
Measure: Count of Participants; unit: Participants
Arm/Group | SURF-201 | Vehicle
Number analyzed (Participants) | 39 | 40
Participants | 35 | 37
Statistical Analysis 1: Comparison: SURF-201 vs Vehicle; Test type: Superiority; p = 0.766, z-test for proportions; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Post-surgical Ocular Pain Score: Number of Participants Achieving an Ocular Pain Score of 0
Description: as for outcome 2
Time Frame: Day 32
Population: Randomized participants who underwent routine uncomplicated cataract surgery and had no missing VAS assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | SURF-201 | Vehicle
Number analyzed (Participants) | 38 | 41
Participants | 35 | 39
Statistical Analysis 1: Comparison: SURF-201 vs Vehicle; Test type: Superiority; p = 0.619, z-test for proportions; [statistical method as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Overall study period
Description: Adverse events were collected from each participant's signature of informed consent at Screening through Day 32 (completion of the study) or early withdrawal.
Arm/Group | SURF-201 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43
Serious Adverse Events (participants affected / at risk) | 3/40 | 0/43
Other Adverse Events (participants affected / at risk) | 26/40 | 23/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SURF-201 (N=40) | Vehicle (N=43)
Cystoid macular edema (Eye disorders) | 1 | 0
Posterior caple rupture (Eye disorders) | 1 | 0
Intraocular pressure increased (Investigations) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SURF-201 (N=40) | Vehicle (N=43)
Visual acuity reduced (Eye disorders) | 6 | 10
Eye inflammation (Eye disorders) | 6 | 8
Posterior capsule opacification (Eye disorders) | 5 | 6
Eye pain (Eye disorders) | 5 | 4
Corneal edema (Eye disorders) | 2 | 4
Photophobia (Eye disorders) | 2 | 3
Conjunctival hyperemia (Eye disorders) | 1 | 3
Iritis (Eye disorders) | 3 | 1
Vitreous detachment (Eye disorders) | 3 | 1
Eye irritation (Eye disorders) | 3 | 0
Vitreous floaters (Eye disorders) | 2 | 1
Intraocular pressure increased (Investigations) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT04324359/Prot_SAP_000.pdf